CLINICAL TRIAL: NCT04000659
Title: A Prospective, Randomized, Controlled, Multi-Center Study to Evaluate the Safety and Effectiveness of the Episealer® Knee System Compared to Microfracture for the Treatment of Focal Femoral Knee Chondral or Osteochondral Lesions
Brief Title: Episealer® Knee System IDE Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Episurf Medical Inc. (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDE 1006
Record Dates: First submitted 2019-06-10; First posted 2019-06-27 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Degenerative Lesion of Articular Cartilage of Knee
Keywords: Knee; Cartilage
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Intervention Model Description: A total of 180 subjects will be enrolled and randomized using a 2:1 ratio (Episealer: Microfracture). Within each site, subjects will be randomized into one of the two study arms using a blocked randomization scheme with varying block sizes.
Who Masked: Participant
Masking Description: In this investigation, neither the investigator nor the subject can be blinded to the treatment group assignment due to the implant's distinctive form that can be detected on radiographs; however, the randomization assignment will not be disclosed to the subject until after surgery is performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Episealer Knee System (Experimental): The experimental arm will comprise of subjects that will be treated with the Episealer Knee System.
  Interventions: Device: Episealer Knee System
- Microfracture (Placebo Comparator): The control arm will comprise of subjects that will receive a Microfracture surgery.
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Device: Episealer Knee System — The Episealer Knee System is comprised of individualized endoprosthetic resurfacing implants and implantation tools (Episealer Toolkit). The implants are designed to replace the articulating surface which has been damaged due to femoral knee chondral and osteochondral defects.
  Arms: Episealer Knee System
Procedure: Microfracture — Microfracture is a minimally invasive surgical technique developed to repair defects in articular cartilage and reduce pain in the knee joint. Microfracture techniques are described in the orthopedic literature and are performed arthroscopically.
  Arms: Microfracture

SUMMARY:
The study is a randomized, prospective, multicenter, controlled clinical trial of the Episealer Knee System. The Episealer Knee System is intended for subjects with up to two focal femoral knee chondral or osteochondral lesion that is causing pain and/or disability and requires surgical treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and clinical effectiveness of the Episealer Knee System (Episealer Trochlea Solo, Episealer Femoral Twin, and Episealer Condyle Solo) compared to microfracture (with or without debridement) in a group of subjects that require repair of up to 2 focal femoral chondral or osteochondral lesions in the knee.

Clinical success will be analyzed via subject reported outcomes to measure function and pain improvements as compared to baseline, incidence of secondary surgical interventions for the treated knee, absence of subsidence or migration through radiographic assessment, and assessment of weight-bearing status.

ELIGIBILITY:
INCLUSION CRITERIA

1. Be ≥ 30 years and ≤ 70 years.
2. Have up to 2 symptomatic femoral chondral or osteochondral defects in the index knee on the medial or lateral femoral condyles or the knee trochlea area, which are:

   1. ICRS Grade 2, 3 or Grade 4
   2. Each suitable for treatment with 1 Episealer device NOTE: Additional femoral cartilage lesions which, in the opinion of the investigator, are asymptomatic and free from underlying bone lesions (e.g., bone edema) will not be treated.
3. Have focal articular defect(s) each with a cartilage lesion area ≥ 1.5 cm2 and ≤ 7.0 cm2.

   1. Subjects with up to two defects ≥ 1.5 cm2 and ≤ 4.0 cm2, that are surrounded by adequate circumferential cartilage as determined by the investigator, will be randomized.
   2. Subjects with at least one defect > 4.0 cm2 and ≤ 7.0 cm2, with adequate bony support as determined by the investigator, will not be randomized, and will receive the Episealer device.
4. Have screening scores that meet the following criteria:

   1. Visual Analog Scale (VAS) pain score of the index knee of ≥ 40 mm
   2. KOOS Overall Score of ≤ 60
5. Have experienced knee pain symptoms and undergone prior non-surgical management (e.g., physical therapy, bracing, HA injections) for at least 4 weeks prior to being considered for the study.
6. Be able to give voluntary, written informed consent to participate and have signed an Informed Consent Form specific to this study.
7. Be willing and able to comply with all study procedures including all pre-operative, post-operative, and rehabilitation requirements.

If female and of child-bearing potential, must have a negative pregnancy test prior to the surgical procedure and no intention of becoming pregnant in the next 24 months.

EXCLUSION CRITERIA

Pre-Operative Exclusion Criteria

Subjects who meet any of the following pre-operative screening criteria will be excluded from participation in this study:

1. Have a Body Mass Index (BMI) greater than 37 kg/m2.
2. Have an ICRS Grade 3 or 4 tibial lesion of any size, or an ICRS Grade 4 patella lesion/fissure ≥ 2.0 mm in width in the index knee.
3. Have malalignment of >8 degrees varus or valgus in the index knee based on standard AP x-rays.
4. Have deficits in flexion or extension of >10 degrees in the index knee as compared to the contralateral knee.
5. Have an existing prosthesis in the index knee compartment or opposing joint surface.
6. Have joint instability in the index knee due to soft tissue or muscular insufficiency.
7. Have a vascular insufficiency at the lesion site that will impair successful microfracture (e.g., avascular necrosis/osteonecrosis, osteochondritis dissecans). (NOTE: This exclusion will not apply to patients with lesions between 4.0-7.0 cm2 who will not undergo randomization and will be treated in the Episealer-only arm).
8. Have inadequate bone stock underlying the lesion site, in the opinion of the investigator.
9. Have any condition, therapy, or medication that may impair bone healing or prevent adequate implant fixation (e.g., osteoporosis).
10. Have a diagnosis of a concomitant knee injury, which in the opinion of the investigator, may confound assessment of the index knee.
11. Have any meniscus tears or defects that require resection of more than 1/3 of the meniscus in the compartment to be treated (i.e., medial meniscus when medial femoral compartment is being treated; lateral meniscus when lateral femoral compartment is being treated).
12. Have a contralateral knee with symptomatic cartilage, meniscal, or ligamentous lesions; generalized osteoarthritis, or any condition that requires surgery, which in the opinion of the investigator, may confound assessment of the index knee, or any condition that requires surgery.
13. Have any condition that is unrelated to the index knee and significantly impairs walking ability (e.g., spinal stenosis, sciatica).
14. Have undergone previous treatment with autograft or allograft transfer, synthetic plugs, or microfracture in the index knee within 6 months of screening. (NOTE: Subjects who have undergone debridement at any point in the past are not excluded).
15. Have a loss of joint space on standing radiographs (Kellgren-Lawrence Grade ≥3) in the index knee.
16. Have an active systemic infection, or an active local infection in or near the index knee, or a previous history of joint infection.
17. Have a history of rheumatoid arthritis.
18. Have known allergies to any of the materials used in the implant (i.e., Cobalt-Chrome alloy and Titanium).
19. Have a contraindication to MRI (e.g., implanted pacemaker, metallic cardiac valve(s), magnetic material such as surgical clips, stent, implanted electronic infusion pumps or any other condition that would prevent the subject from undergoing an MRI).
20. Have a known immunodeficiency including subjects who are receiving or have received corticosteroids, immunosuppressants, immunostimulating agents or radiation therapy within 6 months prior to surgery.
21. Are participating in another clinical investigation for which they received an investigational product (including, but not limited to, a drug or vaccine) within the last 60 days or report the intention to participate in another clinical investigation during the course of the study
22. Are currently abusing drugs or alcohol or have a history of the same within the last 6 months.
23. Have any mental or psychological disorder that would impair their ability to complete the study questionnaires.
24. Are currently breastfeeding or planning to breastfeed any time during the course of the study.
25. Are currently a prisoner.
26. Have significant comorbidities or conditions associated with high-risk for surgical or anesthetic survival (e.g., renal failure, peripheral vascular disease, unstable cardiac disease, poorly controlled diabetes, immunosuppression, etc.).
27. Have any medical condition or other circumstances, in the judgment of the investigator, that might interfere with the ability to return for follow-up visits, including any systemic illness, neuromuscular, neurosensory, or musculoskeletal deficiency that would render the subject unable to perform appropriate post-operative rehabilitation.
28. Have any condition which, in the judgment of the Investigator, would preclude adequate evaluation of the device's safety and performance.

Intra-operative Exclusion Criteria

Subjects who meet any of the following intra-operative screening criteria will be excluded from participation in this study:

1. Have any meniscus tears or defects that require resection of more than 1/3 of the meniscus in the compartment to be treated (i.e., medial meniscus when medial femoral compartment is being treated; lateral meniscus when lateral femoral compartment is being treated).
2. Have chondrosis of the non-operative patellofemoral compartment, contralateral compartment or medial or lateral proximal tibia greater than Outerbridge Grade 2.
3. Have an index lesion on the articular surface that lacks adequate circumferential cartilage as determined by the investigator (NOTE: This exclusion applies only to patients randomized to the microfracture arm.)

   Applicable to Investigational Group Only
4. Have a defect undergoing treatment that cannot be adequately covered by the Episealer device based on intra-operative measurements.

Have bone quality which, in the judgment of the surgeon, would prevent satisfactory fixation of the investigational device.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in the Knee Injury & Osteoarthritis Outcome Score (KOOS) Subscores | 24 Months
  This endpoint will examine the change in KOOS subscores at 24 months
Change in Visual Analog Scale (VAS) Pain Scores | 24 Months
  This endpoint will examine the change in VAS Pain scores at 24 months
Incidence of Secondary Surgical Intervention | 24 Months
  This endpoint will examine the incidence of Secondary Surgical Interventions (SSIs) at 24 months
Incidence of subsidence or migration at 24 months | 24 Months
  This endpoint will examine the incidence of subsidence/migration at 24 months
Weight bearing status | 8 weeks
  This endpoint will examine the weight bearing status at 8 weeks

SECONDARY OUTCOMES:
Change in the KOOS Subscores at all follow-up time points | 3-weeks, 8-weeks, 6-months, 12-months, and 24-months
  This endpoint will examine the change in KOOS subscores at all follow-up time points
Change in VAS Pain score at all follow-up time points | 3-weeks, 8-weeks, 6-months, 12-months, and 24-months
  This endpoint will examine the change in VAS Pain scores at all follow-up time points
Change in 12-Item Short Form Survey (SF-12) score at all follow-up time points | 3-weeks, 8-weeks, 6-months, 12-months, and 24-months
  This endpoint will examine the change in SF-12 scores at all follow-up time points
Incidence of radiographic findings at all follow-up time points | 8 weeks, 12-months, and 24-months
  This endpoint will examine the incidence of radiographic findings at all follow-up time points
Incidence of adverse events and device deficiencies at all follow-up time points | 3-weeks, 8-weeks, 6-months, 12-months and 24-months
  This endpoint will examine the safety via the incidence of adverse events and device deficiencies at all follow-up time points

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Flodström, Study Director — Episurf Medical Inc.
Locations (13):
- United States (8):
  - Physicians Research Group, Tempe, Arizona
  - Horizon Clinical Research, La Mesa, California
  - Ochsner Sports Medicine Institute, New Orleans, Louisiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Plancher Orthopaedics & Sports Medicine, New York, New York
  - Ohio State University, Columbus, Ohio
  - Helios Clinical Research, Jackson, Tennessee
  - North Texas Medical Research Institute, Dallas, Texas
- QEII Health Sciences Center, Halifax, Nova Scotia, Canada
- Germany (2):
  - Universitatsmedizin Berlin Charite, Berlin
  - Orthocentrum Hamburg, Hamburg
- United Kingdom (2):
  - University Hospital Coventry and Warwickshire NHS Trust, Coventry, England
  - University Hospital Southampton NHS Foundation Trust, Southampton, SO16 6YD